CLINICAL TRIAL: NCT06710340
Title: Influence of Acute Nut Intake on the Effects of High Saturated Fat Meals in Obese Diabetic Women
Brief Title: Research on Effects of Acute Consumption of Nuts in Obese Diabetic Women
Acronym: REACT-NUT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Raquel Ballarin (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other)
Responsible Party: Sponsor-Investigator, Raquel Ballarin, Principal Investigator, UPECLIN HC FM Botucatu Unesp
Organization: UPECLIN HC FM Botucatu Unesp (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 80382624.8.0000.5411
Record Dates: First submitted 2024-11-12; First posted 2024-11-29 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Saturated fat-rich meals; Nut intake; Type 2 diabetes; Obesity; Juglans regia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Nuts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nuts in the first meeting (Other): In the first session, after a 10-hour fasting, a high saturated fat meal with 30g of nuts will be offered.
  In the second session, after a 10-hour fasting, a high saturated fat meal without 30g of nuts will be offered.
  Interventions: Dietary Supplement: Nuts in the first meeting
- Nuts in the second meeting (Placebo Comparator): In the first session, after a 10-hour fasting, a high saturated fat meal without 30g of nuts will be offered.
  In the second session, after a 10-hour fasting, a high saturated fat meal with 30g of nuts will be offered.
  Interventions: Other: Nuts in the second meeting

INTERVENTIONS:
Dietary Supplement: Nuts in the first meeting — 30g of walnuts
  Arms: Nuts in the first meeting
Other: Nuts in the second meeting — 30g of walnuts
  Arms: Nuts in the second meeting

SUMMARY:
Obesity is a multifactorial disease in which excess body fat accumulation increases the risk of other chronic diseases such as type 2 diabetes. The primary cause of obesity is the energy imbalance between calories consumed and expended. A balanced diet is essential for weight control and maintaining a healthy body weight. In this context, the intake of a high saturated fat meal (HSFM) plays a detrimental role, contributing to the development of obesity, type 2 diabetes, cancer, cardiovascular diseases, and exacerbating chronic inflammation. Additionally, it may induce metabolic endotoxemia and modulate profiles of circulating microRNAs. Therefore, due to the harmful health impacts of HSFM, studies on metabolomics and circulating microRNA levels could enhance understanding of the mechanisms of walnuts (Juglans regia) in the prevention and treatment of diseases. The aim of this study is to evaluate whether acute walnut supplementation attenuates the inflammatory response, oxidative stress, glycemic response, and regulates the metabolomic and circulating microRNA responses induced by HSFM in women with obesity and type 2 diabetes. The study will be randomized and crossover, including obese, non-insulin-dependent diabetic women aged over 18, without other comorbidities. In the first phase, participants will arrive at the clinic after a 10-hour fast and will be offered HSFM with or without 30g of walnuts. In the second phase, participants who did not receive walnuts will now receive them along with the HSFM and vice versa. Blood samples will be collected, and serum insulin, glucose, serum biomarkers of inflammation and oxidative stress will be evaluated. TNF-alpha, IL-6, IL-1β, IL-1ra, IL-8, and IL-10 will be measured by ELISA, and MDA by HPLC. Additionally, metabolomic and microRNA analyses will be conducted. Data analysis will be performed using JAMOVI v 2.3.21, with a significance level of 5%.

DETAILED DESCRIPTION:
Obesity is a multifactorial disease in which excess body fat accumulation leads to negative health effects. It is considered a global public health problem, primarily due to its association with an increased risk of developing other non-communicable chronic diseases (NCDs). In Brazil, it is estimated that one quarter of the population is obese, making it an important risk factor for pathological aging.

The primary cause of obesity is the energy imbalance between calories consumed and expended, and its high prevalence is associated with physical inactivity and sedentary behavior. A balanced diet, consisting of natural and minimally processed foods, is known to be essential for weight control. However, in the current scenario, there has been a significant increase in the consumption of ultra-processed foods and a decrease in the intake of natural and minimally processed foods, resulting in a major impact on the prevalence of obesity.

Obesity is one of the most relevant risk factors for type 2 diabetes, a disease that is increasingly prevalent worldwide and is considered one of the health emergencies of the 21st century. Diabetes impacts morbidity and mortality and is a major risk factor for stroke, kidney dysfunction, cardiovascular diseases, vision loss, and neuropathy. Non-pharmacological strategies to control diabetes typically include nutritional intervention, regular physical activity, smoking cessation, and maintenance of a healthy body weight.

Acute intake of macronutrients can induce adverse responses even in healthy individuals, which may lead to chronic effects over time. In this context, the intake of a high saturated fat meal (HSFM) plays an important role, as chronic consumption of a HSFM is known to contribute to the development of obesity, type 2 diabetes, cancer, and cardiovascular diseases, as well as exacerbate chronic inflammation induced by insulin resistance and excess weight. Additionally, studies show that HSFM can also induce metabolic endotoxemia and modulate profiles of circulating microRNAs. MicroRNAs are non-coding RNA molecules about 22 nucleotides long that regulate gene expression at the post-transcriptional level by degrading mRNA or inhibiting the translation of target genes. Thus, microRNAs may contribute to the adverse effects of HSFM.

Given the detrimental health impacts of HSFM, studies have been conducted with acute supplementation of foods with anti-inflammatory and antioxidant properties, such as orange juice and green tea, in order to minimize the negative effects of unhealthy diets. A study conducted by our research group showed that acute supplementation of green tea inhibited the expression of 62 microRNAs induced by HSFM intake. Bioinformatics analysis revealed that these microRNAs regulated genes associated with TGF-beta, CARM1, RSK, and BMP pathways. Identifying these miRNAs and their molecular pathways can enhance understanding of the benefits of dietary compounds in health and disease.

Regular walnut consumption (Juglans regia) is associated with better cardiovascular health and insulin response, potentially due to regulation of insulin response by reducing the activity of carbohydrate-digesting enzymes. However, the literature on the effects of walnuts on inflammatory and antioxidant responses remains limited and inconclusive. Furthermore, there is a limited number of studies investigating the acute effects of walnuts, with some evidence of positive responses. In this regard, postprandial attenuation of insulin resistance, improved endothelial function, oxidative stress, and satiety have been demonstrated in some, but not all studies. Interestingly, Torabian et al. observed that acute walnut consumption increased plasma concentrations of polyphenols, enhanced total antioxidant capacity, and reduced plasma lipid peroxidation.

In addition to the limited evidence regarding the acute effects of walnuts, their effects in conjunction with HSFM on metabolomic and microRNA profiles have yet to be studied. Metabolomics was initially defined as the quantitative measurement of the dynamic multiparametric metabolic response of living systems to physiopathological stimuli or genetic modification. Thus, it directly reflects the phenotype of a particular biological system at the molecular metabolic level, allowing for the detection of alterations in previously unknown, uncharacterized, or rarely reported metabolites. Therefore, metabolomics can generate important knowledge about the mechanisms of walnuts in the prevention and treatment of diseases. The same applies to the study of microRNAs, which can assist in identifying intracellular pathways related to the beneficial effects of walnut consumption.

In light of this, this study will generate new evidence regarding the acute effects of walnuts in mitigating the adverse effects of HSFM. Moreover, mitigating the adverse effects of HSFM could yield significant benefits, particularly for patients with insulin resistance, such as the obese and diabetic.

To evaluate whether acute walnut supplementation (Juglans regia) attenuates inflammatory markers, oxidative stress, metabolomics, and circulating microRNAs induced by HSFM in obese and diabetic women.

The project has been approved by the Ethics Committee of the Faculty of Medicine of Botucatu. The study will be randomized and crossover, including women with obesity (body mass index [BMI] ≥ 30) and non-insulin-dependent diabetes aged over 18, recruited during outpatient consultations at the Faculty of Medicine of Botucatu. The exclusion criteria will include: use of dietary supplements, use of corticosteroids in the last 3 months, cancer, heart failure, kidney disease, liver disease, lung disease, neurological diseases, allergy to any component of HSFM or walnuts, and habitual walnut consumption (≤3 times per week) in the past month.

Sample size was estimated based on a previous study that showed a 60% reduction in IL-6 levels after HSFM meals associated with orange juice compared to the control group (without orange juice). Considering this reduction, a type 1 error of 5%, and a power of 90%, this study will include 15 individuals.

Patients who sign the Informed Consent Form (ICF) will be evaluated at two time points, separated by a minimum washout period of one week. In the first meeting, after a 10-hour fast, HSFM will be offered with or without 30g of walnuts. In the second, the condition will be swapped. This walnut dosage refers to the daily consumption recommendation for nuts proposed by various dietary guidelines. Simple randomization will be conducted by a nurse not involved in the research. HSFM will be provided in the hospital outpatient clinic, and patients will be required to consume the entire meal and all the walnuts. During the study protocol, patients will be advised to avoid walnut consumption for 2 weeks prior to the first study visit.

Blood samples will be collected at time points 0 (immediately before the meal), 15 min, 30 min, 60 min, and 150 min after the interventions. Serum insulin and glucose will be measured at time points 0 to 60 min, while serum biomarkers of inflammation, oxidative stress, circulating microRNAs, and metabolomics will be measured at time points 0 and 150 min. Additionally, the investigators will assess satiety using a visual analog scale (VAS) at all time points after the meal.

Metabolomic Analysis The analyses will be conducted using liquid chromatography on a Thermo Dionex Ultimate 3000 system coupled to a high-resolution and accurate mass Thermo QExactive Plus mass spectrometer with electrospray ionization operating in both positive and negative analysis modes.

Analysis of Circulating MicroRNAs After the extraction of RNAs, the investigators will utilize the human miRNA array 4.0 Affymetrix GeneChip® (ThermoFisher Scientific), following the manufacturer's instructions. This array contains 2,578 sets of probes for mature human miRNAs and 2,025 sets of probes for human pre-miRNAs (stem-loop). Probes to detect the presence of snoRNA and scaRNA (a total of 1,996) are also included in this array. The GeneChips will be scanned using the Affymetrix GeneChip G3000 7G scanner, set to capture signal intensities for the miRNAs. The raw intensity data will be imported into the Affymetrix Expression Console (v1.4.1.46) for signal preprocessing, which includes background correction using the robust multi-array average (RMA) algorithm, median polishing summarization of probes to obtain signal values, and quantile normalization across multiple arrays. A detection call for the strength of the miRNA signal will be performed using the Affymetrix "Detection Above Background" (DABG) algorithm, which generates a p-value for each signal above background probability. This method will follow the recommended protocol from the manufacturer. The analyses will be conducted at Monash in Hudson Genomics.

Statistical Analysis Data will be presented as mean and standard deviation when normally distributed, median and 25-75% percentiles when not normally distributed, or as percentages. To compare the two groups (with and without nuts), the investigators will use the Student's t-test for normally distributed data, the Mann-Whitney test for non-normally distributed data, and the Chi-square test for categorical variable comparisons. Additionally, the investigators will apply generalized estimating equations (GEE) to assess repeated measures. Data analyses will be conducted using JAMOVI v 2.3.21, with a significance level set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age
* Diagnosis of obesity (body mass index [BMI >30 kg/m²])
* Diagnosis of non-insulin-dependent type II diabetes

Exclusion Criteria:

* Use of dietary supplements or corticosteroid use in the last 3 months
* Diagnosis of insulin dependent diabetes
* Diagnosis of cancer
* Diagnosis of heart failure
* Diagnosis of kidney diseases
* Diagnosis of liver diseases
* Diagnosis of lung diseases
* Diagnosis ofneurological diseases
* Diagnosis of allergy to any component of the high saturated fat meal or walnuts

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Oxidative stress assessment | 6 weeks
  The cytokines TNF-alpha, IL-6, IL-1β, IL-1ra, IL-8, and IL-10 will be measured by ELISA following the manufacturer's instructions for the kits in pg/mL.
Metabolomic profile assessment | 6 weeks
  Serum concentrations of malondialdehyde (MDA) will be measured by high-performance liquid chromatography (HPLC) based on the reaction with thiobarbituric acid in µmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos M Ferreira, PhD, Principal Investigator — FMB/Unesp
Locations (1):
- São Paulo State University (UNESP), Medical School, Botucatu, Botucatu, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be stored in Excel format on specific folders and backed up on external (USB drive) and cloud storage under the researcher's care. Metadata will include file title, researcher's ORCID, file summary, collection date and project number (if available).
  The project was approved by the Botucatu School of Medicine's Ethics Committee, and informed consent will be obtained from participants or guardians.
  Data will be analyzed in SigmaPlot 12.0, and files will be accessible via standard software. Tabulated data will be preserved indefinitely, with access limited to the research team, and clinical trial data will be anonymized. Tissue samples will be stored at -80°C for up to five years.
  Partial data may be presented at scientific events, and final data will be published as a scientific article. Raw data will be indefinitely retained by the researcher, available upon request, and shared in the institutional repository under anonymization.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study, data will be permanently placed in the institutional repository and made available. Blood samples will be stored in the biorepository for up to five years.
Access Criteria: The data will be available in the institutional repository to anyone upon request.

DOCUMENTS (2):
  • Study Protocol (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT06710340/Prot_000.pdf
  • Informed Consent Form (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT06710340/ICF_001.pdf